CLINICAL TRIAL: NCT01787747
Title: A Phase 1, Single-center, Randomized, Double-blind, Study to Assess the Pharmacokinetics, Safety and Tolerability of Single and Multiple Doses of AVP-786 (Deuterated Dextromethorphan) in Healthy Volunteers
Brief Title: Pharmacokinetics (PK) and Tolerability of AVP-786 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 12-AVR-132
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Healthy Volunteers; dextromethorphan with quinidine; deuterated dextromethorphan
MeSH Terms: interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohorts A and C (Experimental): Single dose (D1) followed by twice daily dosing for 7 days
  Interventions: Drug: AVP-786 Dose 1; Drug: AVP-923
- Cohorts B and D (Experimental): Single dose (D1) followed by twice daily dosing for 7 days
  Interventions: Drug: AVP-786 Dose 2; Drug: AVP-923
- Cohorts E and F (Experimental): Single dose (D1) followed by twice daily dosing for 7 days
  Interventions: Drug: AVP-786 Dose 1/Q Dose 1; Drug: AVP-923
- Cohorts G and I (Experimental): Single dose (D1) followed by twice daily dosing for 7 days
  Interventions: Drug: AVP-786 Dose 1/Q Dose 2; Drug: AVP-923
- Cohorts H and J (Experimental): Single dose (D1) followed by twice daily dosing for 7 days
  Interventions: Drug: AVP-786 Dose 2/Q Dose 2; Drug: AVP-923

INTERVENTIONS:
Drug: AVP-786 Dose 1
  Arms: Cohorts A and C
Drug: AVP-786 Dose 2
  Arms: Cohorts B and D
Drug: AVP-786 Dose 1/Q Dose 1
  Arms: Cohorts E and F
Drug: AVP-786 Dose 1/Q Dose 2
  Arms: Cohorts G and I
Drug: AVP-786 Dose 2/Q Dose 2
  Arms: Cohorts H and J
Drug: AVP-923

SUMMARY:
To assess the single- and multiple-dose pharmacokinetic (PK), safety and tolerability of AVP-786 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males
* 18 - 45 years of age
* BMI 18 - 30 kg/m2

Exclusion Criteria:

* History or presence of significant disease
* History of substance and/or alcohol abuse within the past 3 years
* Use of tobacco-containing or nicotine-contining products within 6 months
* Use of any prescription of over-the-counter (OTC) medication within 14 days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of parent and metabolites | 8 Days

SECONDARY OUTCOMES:
Safety and tolerability | 8 days
  Assessments to include Physical Examination (PE), Labs, ECGs, and Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — CMAX
Locations (1):
- CMAX, Adelaide, South Australia, Australia